CLINICAL TRIAL: NCT01334840
Title: Mechanism of Action of Vichy Catalan Water
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Vichy Catalán, Spain (Unknown)
Responsible Party: M Pilar Vaquero, National Research Council, Spain
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: BW-09
Record Dates: First submitted 2011-04-12; First posted 2011-04-13 (Estimated); Last update posted 2014-07-30 (Estimated); Status verified 2011-04

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular risk; Cholecystokinin; Gallbladder emptying; Lipid absorption; Postprandial triacylglycerols; Sodium-bicarbonated mineral water
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (4):
- BW (Experimental): Bicarbonated mineral water without meal
  Interventions: Dietary Supplement: Bicarbonated mineral water
- BW with meal (Experimental): Bicarbonated mineral water with meal
  Interventions: Dietary Supplement: Bicarbonated mineral water
- CW (Active Comparator): Mineral water low in mineral content (control) without meal
  Interventions: Dietary Supplement: Mineral water low in mineral content (control)
- CW with meal (Active Comparator): Mineral water low in mineral content (control) with a meal
  Interventions: Dietary Supplement: Mineral water low in mineral content (control)

INTERVENTIONS:
Dietary Supplement: Bicarbonated mineral water — Volunteers fasted overnight consumed:
  0.5 L of the bicarbonated mineral water without meal or, 0.5 L of the bicarbonated mineral water with meal
  Arms: BW; BW with meal
Dietary Supplement: Mineral water low in mineral content (control) — Volunteers fasted overnight consumed:
  0.5 L of the control water without meal or, 0.5 L of the control water with meal
  Arms: CW; CW with meal

SUMMARY:
Water consumption is essential to maintain hydration and good health. Sodium-bicarbonated mineral waters are reported to have beneficial digestive and hypocholesterolemic properties. The aim of this study was to investigate the effects of the consumption of a sodium-bicarbonated mineral water (BW) with or without a meal, compared to a low mineral content water as a control water (CW), on postprandial serum triacylglycerols (TAG), cholecystokinin (CCK), and gallbladder volume.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 and <40 years)
* BMI >18 and <30 kg/m2

Exclusion Criteria:

* Age <18 and > 40 years
* TAG > 250 mg/dL (2.82 mmol/L)
* Being a usual consumer of carbonic mineral water
* Obesity
* Diabetes
* Hypertension or digestive, liver and renal disease
* Biliary obstruction
* Eating disorders
* Being under medication that could affect lipid metabolism
* Consumption of functional foods that could affect lipid metabolism (food containing n-3 fatty acids or phytosterols)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Serum triacylglycerols | Baseline
Serum triacylglycerols | Postprandial 30 minutes
Serum triacylglycerols | Postprandial 60 minutes
Serum triacylglycerols | Postprandial 120 minutes

SECONDARY OUTCOMES:
Serum glucose | Baseline
Serum glucose | Postprandial 30 minutes
Serum glucose | Postprandial time 60 minutes
Serum glucose | Postprandial time 120 minutes
Serum insulin | Baseline
Serum insulin | Postprandial 30 minutes
Serum insulin | Postprandial 60 minutes
Serum insulin | Postprandial 120 minutes
Cholecystokinin | Baseline
Cholecystokinin | Postprandial 30 minutes
Cholecystokinin | Postprandial 60 minutes
Cholecystokinin | Postprandial 120 minutes
Gallbladder volume | Baseline
Gallbladder volume | Postprandial 15 minutes
Gallbladder volume | Postprandial 30 minutes
Gallbladder volume | Postprandial 60 minutes
Gallbladder volume | Postprandial 120 minutes
Aldosterone | Baseline
Aldosterone | Postprandial 30 minutes
Aldosterone | Postprandial 60 minutes
Aldosterone | Postprandial 120 minutes

CONTACTS AND LOCATIONS:
Overall Officials: M Pilar Vaquero, Dr, Principal Investigator — National Research Council, Spain
Locations (1):
- Institute of Food Science, Technology and Nutrition (ICTAN), Spanish National Research Council (CISC), Madrid, Madrid, Spain

REFERENCES:
- [Background] Schoppen S, Perez-Granados AM, Carbajal A, Oubina P, Sanchez-Muniz FJ, Gomez-Gerique JA, Vaquero MP. A sodium-rich carbonated mineral water reduces cardiovascular risk in postmenopausal women. J Nutr. 2004 May;134(5):1058-63. doi: 10.1093/jn/134.5.1058. PMID 15113945
- [Background] Schoppen S, Perez-Granados AM, Carbajal A, de la Piedra C, Pilar Vaquero M. Bone remodelling is not affected by consumption of a sodium-rich carbonated mineral water in healthy postmenopausal women. Br J Nutr. 2005 Mar;93(3):339-44. doi: 10.1079/bjn20041332. PMID 15877873
- [Background] Schoppen S, Perez-Granados AM, Carbajal A, Sarria B, Sanchez-Muniz FJ, Gomez-Gerique JA, Pilar Vaquero M. Sodium bicarbonated mineral water decreases postprandial lipaemia in postmenopausal women compared to a low mineral water. Br J Nutr. 2005 Oct;94(4):582-7. doi: 10.1079/bjn20051515. PMID 16197584
- [Background] Schoppen S, Perez-Granados AM, Carbajal A, Sarria B, Navas-Carretero S, Pilar Vaquero M. Sodium-bicarbonated mineral water decreases aldosterone levels without affecting urinary excretion of bone minerals. Int J Food Sci Nutr. 2008 Jun;59(4):347-55. doi: 10.1080/09637480701560308. PMID 17886090
- [Background] Schoppen S, Sanchez-Muniz FJ, Perez-Granados M, Gomez-Gerique JA, Sarria B, Navas-Carretero S, Pilar Vaquero M. Does bicarbonated mineral water rich in sodium change insulin sensitivity of postmenopausal women? Nutr Hosp. 2007 Sep-Oct;22(5):538-44. PMID 17970536
- [Background] Perez-Granados AM, Navas-Carretero S, Schoppen S, Vaquero MP. Reduction in cardiovascular risk by sodium-bicarbonated mineral water in moderately hypercholesterolemic young adults. J Nutr Biochem. 2010 Oct;21(10):948-53. doi: 10.1016/j.jnutbio.2009.07.010. Epub 2009 Dec 1. PMID 19954956
- [Background] Schoppen S, Perez-Granados AM, Navas-Carretero S, Vaquero MP. Postprandial lipaemia and endothelial adhesion molecules in pre- and postmenopausal Spanish women. Nutr Hosp. 2010 Mar-Apr;25(2):256-61. PMID 20449535
- [Result] Toxqui L, Perez-Granados AM, Blanco-Rojo R, Vaquero MP. A sodium-bicarbonated mineral water reduces gallbladder emptying and postprandial lipaemia: a randomised four-way crossover study. Eur J Nutr. 2012 Aug;51(5):607-14. doi: 10.1007/s00394-011-0244-x. Epub 2011 Sep 13. PMID 21913027
- [Result] Toxqui L, Pérez-Granados AM, Blanco-Rojo R, Vaquero MP. Effects of an alkaline mineral water on cholecystokinin levels and gallbladder emptying in young adults. Ann Nutr Metab 58(suppl 3):352-353,2011
- [Result] Toxqui L, Pérez-Granados AM, Blanco-Rojo R, Vaquero MP. Sodium-bicarbonated mineral water reduces postprandial lipaemia in moderately hypercholesterolaemic young adults. Proceedings of the Nutrition Society 70 (OCE4):E245, 2011.
- [Derived] Toxqui L, Vaquero MP. Aldosterone changes after consumption of a sodium-bicarbonated mineral water in humans. A four-way randomized controlled trial. J Physiol Biochem. 2016 Dec;72(4):635-641. doi: 10.1007/s13105-016-0502-8. Epub 2016 Jun 29. PMID 27356528